CLINICAL TRIAL: NCT07402083
Title: Administration of Extracellular Vesicles Isolated From Donor Human Milk as a Dietary Supplement for the Prevention of Necrotizing Enterocolitis in Preterm Infants
Brief Title: Administration of Extracellular Vesicles From Donor Human Milk in Preterm Infants
Acronym: AdVEMPrem
Status: Recruiting | Type: Observational
Sponsor: Instituto de Investigacion Sanitaria La Fe (Other)
Collaborators: Hospital Universitario La Fe (Other)
Responsible Party: Sponsor
Other Study IDs: PI23/00202; PI23/00202 (Other: Instituto de Salud Carlos III (ISCIII))
Record Dates: First submitted 2025-12-09; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Very Preterm Infants (<32 Weeks of Gestation)
Keywords: Preterm birth (<32 weeks); Donor human milk (DHM); Extracellular vesicles (EVs); Feeding tolerance; Necrotizing enterocolitis (NEC); Neurodevelopment; Donor Human Milk Extracellular Vesicle (DHMEVs)
MeSH Terms: conditions — Premature Birth; Enterocolitis, Necrotizing

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The study will retain biological samples collected from preterm infants, own mother's milk (OMM), and donor human milk (DHM) to support biochemical and functional analyses. Specifically:
  1. OMM/DHM samples: isolation of extracellular vesicles (EVs), lipid profiling, and compositional characterization, and functional assays.
  2. Infant urine samples: redox status and oxidative/nitrosative stress biomarkers.
  3. Maternal urine samples: food intake biomarkers.
  4. Infant blood samples (minimally invasive micro-sampling, e.g., dried blood spots and plasma samples): redox status (oxidized/reduced glutathione) and inflammation biomarker determination.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- EV supplementation in very preterm infants: Infants born before 32 weeks of gestation will receive own mother's milk supplemented with extracellular vesicles isolated from donor human milk.
  Interventions: Dietary Supplement: Donor human milk extracellular vesicles (DHM-EVs)

INTERVENTIONS:
Dietary Supplement: Donor human milk extracellular vesicles (DHM-EVs) — Infants born before 32 weeks of gestation will receive supplementation with extracellular vesicles isolated from donor human milk, in addition to standard nutritional care.

SUMMARY:
The AdVEMPrem study is exploring whether tiny particles called extracellular vesicles (EVs), which are naturally found in human milk, can help protect very premature babies from serious gut problems such as necrotizing enterocolitis (NEC). NEC is a dangerous condition that affects the intestines of preterm infants and can lead to long-term health issues.

Human milk is the best nutrition for babies, but when a mother's own milk is not available, donor human milk (DHM) is used. EVs in milk carry proteins, fats, and genetic material that may support gut development, immunity, and brain growth. While laboratory studies suggest EVs are beneficial, their effects in premature babies have not yet been proven.

In this study, 20 very preterm infants (<32 weeks of gestation) will be enrolled during their stay in the Neonatal Intensive Care Unit (NICU). All babies in the study will receive oral supplementation with EVs isolated from donor human milk. Researchers will monitor feeding tolerance, growth, intestinal health, and early development. Blood and urine samples will also be collected to study how EVs affect metabolism and stress markers.

The main goal is to see if EV supplementation is safe and well tolerated. Longer-term follow-up will explore whether EVs improve growth and neurodevelopment as the babies grow. This research could lead to new nutritional strategies to reduce NEC and improve outcomes for premature infants and their families.

DETAILED DESCRIPTION:
Human milk is the optimal source of nutrition for infants, providing essential nutrients and bioactive components that promote growth and development. Very preterm infants (<32 weeks gestation) are particularly vulnerable to feeding intolerance, impaired growth, and severe complications such as necrotizing enterocolitis (NEC). When a mother's own milk is insufficient or unavailable, pasteurized donor human milk (DHM) is the recommended alternative.

Extracellular vesicles (EVs) are nanosized particles naturally present in human milk that carry proteins, lipids, and nucleic acids involved in cell signaling, intestinal maturation, immune regulation, and neurodevelopment. Preclinical studies suggest that milk-derived EVs may reduce inflammation and support gut and brain development, but their role in clinical outcomes for very preterm infants has not yet been established.

The AdVEMPrem study (PI23/00202, ISCIII) is a prospective, single-arm pilot trial designed to evaluate the tolerance and safety of DHM-derived EV supplementation in very preterm infants. All enrolled infants will receive oral EV supplementation during hospitalization in the Neonatal Intensive Care Unit. Protocols for isolation and quality control of DHM-EVs will be established to ensure reproducible yields. The biochemical composition of milk and EVs will be characterized for product characterization and exploratory analyses, with emphasis on lipid profiles and functional properties. These analyses are not participant-level outcome measures. Clinical, nutritional, and developmental parameters will be monitored during the neonatal period, alongside biomarkers of redox balance and oxidative/nitrosative stress. Long-term follow-up will assess sustained effects on growth and neurodevelopmental trajectories.

Findings from this pilot study will provide foundational evidence for the potential of milk-derived EVs as a safe nutritional strategy to prevent NEC and improve outcomes in preterm infants. Results will inform the design of larger multicenter trials and may contribute to the development of standardized EV-based supplements or analogues from alternative sources, thereby addressing variability in donor milk composition. Ultimately, access to an efficient and safe nutritional supplement could reduce the incidence of NEC, improve infant and family outcomes, and deliver socio-economic and ecological benefits.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants born at <32 weeks gestational age
* Age between 0 and 14 days of life at enrollment
* At risk of developing necrotizing enterocolitis (NEC)
* Written informed consent obtained from parent(s) or legal guardian(s)

Exclusion Criteria:

* Major congenital anomalies or chromosomal abnormalities
* Severe gastrointestinal malformations (e.g., gastroschisis, intestinal atresia)
* Conditions incompatible with enteral feeding or EV supplementation
* Participation in another interventional clinical trial

Ages: 0 Days to 14 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Preterm infants at risk of developing necrotizing enterocolitis (NEC), recruited between 14 and 28 days of life during their stay in the Neonatal Intensive Care Unit (NICU). A total of 20 infants will be enrolled to receive oral administration of extracellular vesicles (EVs) isolated from donor human milk (DHM) as a dietary supplement.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2026-02-05 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related serious adverse events | From enrollment until term-equivalent age (i.e., up to 40 weeks postmenstrual age)
  Safety will be evaluated by the number of participants experiencing one or more treatment-related serious adverse events, defined as any of the following: (i) necrotizing enterocolitis (Bell stage ≥ II); (ii) metabolic or renal complications requiring medical intervention, (iii) cholestasis, or (iv) culture-proven sepsis. Participants experiencing multiple events will be counted once.
Tolerance of donor human milk EV supplementation | From enrollment until term-equivalent age (i.e., up to 40 weeks postmenstrual age)
  Feeding tolerance is evaluated by the number of participants without clinical signs of gastrointestinal symptoms and successful progression of enteral feeding.

SECONDARY OUTCOMES:
Infant weight | From enrollment until term-equivalent age (weekly) and at 3, 6, 12, 18, and 24 months of corrected age
  Measurements of weight (grams)
Infant length | From enrollment until term-equivalent age (weekly) and at 3, 6, 12, 18, and 24 months of corrected age
  Measurements of length (cm)
Infant head circumference | From enrollment until term-equivalent age (weekly) and at 3, 6, 12, 18, and 24 months of corrected age
  Measurement of head circumference (cm)
Analysis of redox status biomarkers | 21 days of life
  Evaluation of the ratio reduced/oxidized glutathione
Concentration of TFN alpha (inflammatory biomarker) | 21 days of life
  Evaluation of TFN alpha in plasma employing an Enzyme-Linked Immunosorbent Assay (ELISA) kit (nM)
Concentration of IL-6 (inflammatory biomarker) | 21 days of life
  Evaluation of IL-6 in plasma employing an ELISA kit (nM)
Concentration of calprotectin (inflammation biomarker) | 21 days of life
  Evaluation of calprotectin in plasma employing an ELISA kit (nM)
Ratio of meta-tyrosine/phenylalanine | 14, 21, and 28 days of life
  Evaluation of the ratio of meta-tyrosine/phenylalanine in urine samples by Liquid Chromatography coupled to tandem Mass Spectrometry (LC-MS/MS) as an indicator of oxidative damage to proteins
Ratio of ortho-tyrosine/phenylalanine | 14, 21, and 28 days of life
  Evaluation of the ratio of ortho-tyrosine/phenylalanine in urine samples by LC-MS/MS as an indicator of oxidative damage to proteins
Ratio of 8-hydroxy-2'-deoxyguanosine/2'-deoxyguanosine | 14, 21, and 28 days of life
  Evaluation of the ratio of 8-hydroxy-2'-deoxyguanosine/2'-deoxyguanosine in urine samples by LC-MS/MS as an indicator of oxidative damage to DNA
Concentrations of 2,3-dinor-iPF2α-III | 14, 21, and 28 days of life
  Evaluation of 2,3-dinor-iPF2α-III in urine samples by LC-MS/MS as an indicator of oxidative damage to lipids (n mol/g creatinine)
Concentrations of 5-iPF2α-VI | 14, 21, and 28 days of life
  Evaluation of 5-iPF2α-VI in urine samples by LC-MS/MS as an indicator of oxidative damage to lipids (n mol/g creatinine)
Bayley Scales of Infant and Toddler Development, Fourth Edition (Bayley-IV) - Motor Composite Score | 6 and 24 months corrected age
  Motor development will be assessed using the Motor Composite Score of the Bayley-IV. Higher scores indicate better motor development.
Bayley Scales of Infant and Toddler Development, Fourth Edition (Bayley-IV) Language Composite Score | 6 and 24 months corrected age
  Language development will be assessed using the Language Composite Score of the Bayley-IV. Higher scores indicate better language development.
Bayley Scales of Infant and Toddler Development, Fourth Edition (Bayley-IV) - Cognitive Composite Score | 6 and 24 months of corrected age
  Neurodevelopment will be assessed using the Cognitive Composite Score of the Bayley Scales of Infant and Toddler Development, Fourth Edition (Bayley-IV). Higher scores indicate better cognitive development.
Ages and Stages Questionnaire, Third Edition (ASQ-3) Total Score | 6 and 24 months of corrected age
  Developmental screening will be assessed using the Ages and Stages Questionnaire, Third Edition (ASQ-3). The ASQ-3 is a parent-completed developmental screening tool consisting of five domains (communication, gross motor, fine motor, problem solving, and personal-social skills). Higher scores indicating better overall development.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario y Politécnico La Fe, Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Albiach-Delgado A, Pinilla-Gonzalez A, Cascant-Vilaplana MM, Solaz-Garcia A, Torrejon-Rodriguez L, Lara-Canton I, Parra-Llorca A, Cernada M, Gormaz M, Pertierra A, Tapia C, Iriondo M, Aguar M, Kuligowski J, Vento M. The effect of inhaled nitric oxide treatment on biomarkers of oxidative/nitrosative damage to proteins and DNA/RNA. Free Radic Biol Med. 2025 Feb 16;228:350-359. doi: 10.1016/j.freeradbiomed.2025.01.020. Epub 2025 Jan 14. PMID 39818239
- [Background] Ramos-Garcia V, Ten-Doménech I, Moreno-Giménez A, Gormaz M, Parra-Llorca A, Shephard AP, et al. ATR-FTIR spectroscopy for the routine quality control of exosome isolations. Chemometrics and Intelligent Laboratory Systems 2021:104401. https://doi.org/10.1016/j.chemolab.2021.104401.
- [Background] Buratta S, Urbanelli L, Tognoloni A, Latella R, Cerrotti G, Emiliani C, et al. Protein and Lipid Content of Milk Extracellular Vesicles: A Comparative Overview. Life 2023;13:401. https://doi.org/10.3390/life13020401.
- [Background] Pisano C, Galley J, Elbahrawy M, Wang Y, Farrell A, Brigstock D, et al. Human Breast Milk-Derived Extracellular Vesicles in the Protection Against Experimental Necrotizing Enterocolitis. Journal of Pediatric Surgery 2020;55:54 -8. https://doi.org/10.1016/j. jpedsurg.2019.09.052.
- [Background] Miyake H, Lee C, Chusilp S, Bhalla M, Li B, Pitino M, et al. Human breast milk exosomes attenuate intestinal damage. Pediatr
- [Background] Liao Y, Du X, Li J, Lönnerdal B. Human milk exosomes and their microRNAs survive digestion in vitro and are taken up by human intestinal cells. Molecular Nutrition & Food Research 2017;61:1700082. https://doi.org/10.1002/mnfr.201700082.
- [Background] Galley JD, Besner GE. The Therapeutic Potential of Breast Milk-Derived Extracellular Vesicles. Nutrients. 2020 Mar 11;12(3):745. doi: 10.3390/nu12030745. PMID 32168961
- [Background] Chutipongtanate S, Morrow AL, Newburg DS. Human Milk Extracellular Vesicles: A Biological System with Clinical Implications. Cells. 2022 Jul 30;11(15):2345. doi: 10.3390/cells11152345. PMID 35954189
- [Background] Lonnerdal B. Human Milk MicroRNAs/Exosomes: Composition and Biological Effects. Nestle Nutr Inst Workshop Ser. 2019;90:83-92. doi: 10.1159/000490297. Epub 2019 Mar 13. PMID 30865991
- [Background] Chen W, Chen X, Qian Y, Wang X, Zhou Y, Yan X, et al. Lipidomic Profiling of Human Milk Derived Exosomes and Their Emerging Roles in the Prevention of Necrotizing Enterocolitis. Mol Nutr Food Res 2021;65:e2000845. https://doi.org/10.1002/ mnfr.202000845.
- [Background] Zonneveld MI, Brisson AR, van Herwijnen MJC, Tan S, van de Lest CHA, Redegeld FA, et al. Recovery of extracellular vesicles from human breast milk is influenced by sample collection and vesicle isolation procedures. J Extracell Vesicles 2014;3. https://doi. org/10.3402/jev.v3.24215.
- [Background] Admyre C, Johansson SM, Qazi KR, Filén J-J, Lahesmaa R, Norman M, et al. Exosomes with immune modulatory features are present in human breast milk. J Immunol 2007;179:1969 -78. https://doi.org/10.4049/jimmunol.179.3.1969.
- [Background] Thery C, Witwer KW, Aikawa E, Alcaraz MJ, Anderson JD, Andriantsitohaina R, Antoniou A, Arab T, Archer F, Atkin-Smith GK, Ayre DC, Bach JM, Bachurski D, Baharvand H, Balaj L, Baldacchino S, Bauer NN, Baxter AA, Bebawy M, Beckham C, Bedina Zavec A, Benmoussa A, Berardi AC, Bergese P, Bielska E, Blenkiron C, Bobis-Wozowicz S, Boilard E, Boireau W, Bongiovanni A, Borras FE, Bosch S, Boulanger CM, Breakefield X, Breglio AM, Brennan MA, Brigstock DR, Brisson A, Broekman ML, Bromberg JF, Bryl-Gorecka P, Buch S, Buck AH, Burger D, Busatto S, Buschmann D, Bussolati B, Buzas EI, Byrd JB, Camussi G, Carter DR, Caruso S, Chamley LW, Chang YT, Chen C, Chen S, Cheng L, Chin AR, Clayton A, Clerici SP, Cocks A, Cocucci E, Coffey RJ, Cordeiro-da-Silva A, Couch Y, Coumans FA, Coyle B, Crescitelli R, Criado MF, D'Souza-Schorey C, Das S, Datta Chaudhuri A, de Candia P, De Santana EF, De Wever O, Del Portillo HA, Demaret T, Deville S, Devitt A, Dhondt B, Di Vizio D, Dieterich LC, Dolo V, Dominguez Rubio AP, Dominici M, Dourado MR, Driedonks TA, Duarte FV, Duncan HM, Eichenberger RM, Ekstrom K, El Andaloussi S, Elie-Caille C, Erdbrugger U, Falcon-Perez JM, Fatima F, Fish JE, Flores-Bellver M, Forsonits A, Frelet-Barrand A, Fricke F, Fuhrmann G, Gabrielsson S, Gamez-Valero A, Gardiner C, Gartner K, Gaudin R, Gho YS, Giebel B, Gilbert C, Gimona M, Giusti I, Goberdhan DC, Gorgens A, Gorski SM, Greening DW, Gross JC, Gualerzi A, Gupta GN, Gustafson D, Handberg A, Haraszti RA, Harrison P, Hegyesi H, Hendrix A, Hill AF, Hochberg FH, Hoffmann KF, Holder B, Holthofer H, Hosseinkhani B, Hu G, Huang Y, Huber V, Hunt S, Ibrahim AG, Ikezu T, Inal JM, Isin M, Ivanova A, Jackson HK, Jacobsen S, Jay SM, Jayachandran M, Jenster G, Jiang L, Johnson SM, Jones JC, Jong A, Jovanovic-Talisman T, Jung S, Kalluri R, Kano SI, Kaur S, Kawamura Y, Keller ET, Khamari D, Khomyakova E, Khvorova A, Kierulf P, Kim KP, Kislinger T, Klingeborn M, Klinke DJ 2nd, Kornek M, Kosanovic MM, Kovacs AF, Kramer-Albers EM, Krasemann S, Krause M, Kurochkin IV, Kusuma GD, Kuypers S, Laitinen S, Langevin SM, Languino LR, Lannigan J, Lasser C, Laurent LC, Lavieu G, Lazaro-Ibanez E, Le Lay S, Lee MS, Lee YXF, Lemos DS, Lenassi M, Leszczynska A, Li IT, Liao K, Libregts SF, Ligeti E, Lim R, Lim SK, Line A, Linnemannstons K, Llorente A, Lombard CA, Lorenowicz MJ, Lorincz AM, Lotvall J, Lovett J, Lowry MC, Loyer X, Lu Q, Lukomska B, Lunavat TR, Maas SL, Malhi H, Marcilla A, Mariani J, Mariscal J, Martens-Uzunova ES, Martin-Jaular L, Martinez MC, Martins VR, Mathieu M, Mathivanan S, Maugeri M, McGinnis LK, McVey MJ, Meckes DG Jr, Meehan KL, Mertens I, Minciacchi VR, Moller A, Moller Jorgensen M, Morales-Kastresana A, Morhayim J, Mullier F, Muraca M, Musante L, Mussack V, Muth DC, Myburgh KH, Najrana T, Nawaz M, Nazarenko I, Nejsum P, Neri C, Neri T, Nieuwland R, Nimrichter L, Nolan JP, Nolte-'t Hoen EN, Noren Hooten N, O'Driscoll L, O'Grady T, O'Loghlen A, Ochiya T, Olivier M, Ortiz A, Ortiz LA, Osteikoetxea X, Ostergaard O, Ostrowski M, Park J, Pegtel DM, Peinado H, Perut F, Pfaffl MW, Phinney DG, Pieters BC, Pink RC, Pisetsky DS, Pogge von Strandmann E, Polakovicova I, Poon IK, Powell BH, Prada I, Pulliam L, Quesenberry P, Radeghieri A, Raffai RL, Raimondo S, Rak J, Ramirez MI, Raposo G, Rayyan MS, Regev-Rudzki N, Ricklefs FL, Robbins PD, Roberts DD, Rodrigues SC, Rohde E, Rome S, Rouschop KM, Rughetti A, Russell AE, Saa P, Sahoo S, Salas-Huenuleo E, Sanchez C, Saugstad JA, Saul MJ, Schiffelers RM, Schneider R, Schoyen TH, Scott A, Shahaj E, Sharma S, Shatnyeva O, Shekari F, Shelke GV, Shetty AK, Shiba K, Siljander PR, Silva AM, Skowronek A, Snyder OL 2nd, Soares RP, Sodar BW, Soekmadji C, Sotillo J, Stahl PD, Stoorvogel W, Stott SL, Strasser EF, Swift S, Tahara H, Tewari M, Timms K, Tiwari S, Tixeira R, Tkach M, Toh WS, Tomasini R, Torrecilhas AC, Tosar JP, Toxavidis V, Urbanelli L, Vader P, van Balkom BW, van der Grein SG, Van Deun J, van Herwijnen MJ, Van Keuren-Jensen K, van Niel G, van Royen ME, van Wijnen AJ, Vasconcelos MH, Vechetti IJ Jr, Veit TD, Vella LJ, Velot E, Verweij FJ, Vestad B, Vinas JL, Visnovitz T, Vukman KV, Wahlgren J, Watson DC, Wauben MH, Weaver A, Webber JP, Weber V, Wehman AM, Weiss DJ, Welsh JA, Wendt S, Wheelock AM, Wiener Z, Witte L, Wolfram J, Xagorari A, Xander P, Xu J, Yan X, Yanez-Mo M, Yin H, Yuana Y, Zappulli V, Zarubova J, Zekas V, Zhang JY, Zhao Z, Zheng L, Zheutlin AR, Zickler AM, Zimmermann P, Zivkovic AM, Zocco D, Zuba-Surma EK. Minimal information for studies of extracellular vesicles 2018 (MISEV2018): a position statement of the International Society for Extracellular Vesicles and update of the MISEV2014 guidelines. J Extracell Vesicles. 2018 Nov 23;7(1):1535750. doi: 10.1080/20013078.2018.1535750. eCollection 2018. PMID 30637094
- [Background] Colombo M, Raposo G, Thery C. Biogenesis, secretion, and intercellular interactions of exosomes and other extracellular vesicles. Annu Rev Cell Dev Biol. 2014;30:255-89. doi: 10.1146/annurev-cellbio-101512-122326. Epub 2014 Aug 21. PMID 25288114
- [Background] Ascanius SR, Hansen MS, Ostenfeld MS, Rasmussen JT. Milk-Derived Extracellular Vesicles Suppress Inflammatory Cytokine Expression and Nuclear Factor-κB Activation in Lipopolysaccharide-Stimulated Macrophages. Dairy 2021;2:165 -78. https://doi. org/10.3390/dairy2020015.
- [Background] Meng F, Uniacke-Lowe T, Ryan AC, Kelly AL. The composition and physico-chemical properties of human milk: A review. Trends in Food Science & Technology 2021;112:608 -21. https://doi.org/10.1016/j.tifs.2021.03.040.
- [Background] Flahive C, Schlegel A, Mezoff EA. Necrotizing Enterocolitis: Updates on Morbidity and Mortality Outcomes. J Pediatr. 2020 May;220:7-9. doi: 10.1016/j.jpeds.2019.12.035. Epub 2020 Jan 16. No abstract available. PMID 31955884
- [Background] Poulimeneas D, Bathrellou E, Antonogeorgos G, Mamalaki E, Kouvari M, Kuligowski J, et al. Feeding the preterm infant: an overview of the evidence. Int J Food Sci Nutr 2021;72:4 -13. https://doi.org/10.1080/09637486.2020.1754352.
- [Background] Garcia C, Duan RD, Brévaut-Malaty V, Gire C, Millet V, Simeoni U, et al. Bioactive compounds in human milk and intestinal health and maturity in preterm newborn: an overview. Cell Mol Biol (Noisy-Le-Grand) 2013;59:108 -31.
- [Result] Method for Mid-IR Spectroscopy of Extracellular Vesicles at the Subvesicle Level, Nikolaus Hondl, Lena Neubauer, Victoria Ramos-Garcia, Julia Kuligowski, Marina Bishara, Eva Sevcsik, Bernhard Lendl, Georg Ramer, ACS Measurement Science Au, DOI: 10.1021/acsmeasuresciau.5c00001
- [Result] Simultaneous Screening and Quantitation of Human Milk Oligosaccharides by Liquid Chromatography - Mass Spectrometry, Víctor Navarro-Esteve, Anna Zöchner, Marta Roca, Anna Parra-Llorca, Alba Moreno-Giménez, Laura Campos-Berga, María Jesús Vaya, Máximo Vento, Pilar Sáenz-González, María Gormaz, Isabel Ten-Domenech, Julia Kuligowski, Guillermo Quintás, Carbohydrate Polymer Technologies and Applications 9 (2024) 100644. doi: 10.1016/j.carpta.2024.100644
- [Result] Normalization approaches for extracellular vesicle-derived lipidomic fingerprints - A human milk case study, Isabel Ten-Doménech, Victoria Ramos-Garcia, Abel Albiach- Delgado, Jose Luis Moreno-Casillas, Alba Moreno-Giménez, María Gormaz, Marta Gómez-Ferrer, Pilar Sepúlveda, Máximo Vento, Guillermo Quintás, Julia Kuligowski, Chemometrics and Intelligent Laboratory Systems 246 (2024) 105070. doi: https://doi.org/10.1016/j.chemolab.2024.105070
- [Result] Ten-Domenech I, Moreno-Gimenez A, Campos-Berga L, Zapata de Miguel C, Lopez-Nogueroles M, Parra-Llorca A, Quintas G, Garcia-Blanco A, Gormaz M, Kuligowski J. Impact of maternal health and stress on steroid hormone profiles in human milk: Implications for infant development. J Lipid Res. 2024 Dec;65(12):100688. doi: 10.1016/j.jlr.2024.100688. Epub 2024 Oct 26. PMID 39490927
- [Result] Kuligowski J, Moreno-Torres M, Quintas G. Improving insights from metabolomic functional analysis combining multivariate tools. Anal Chim Acta. 2024 Sep 22;1323:343062. doi: 10.1016/j.aca.2024.343062. Epub 2024 Aug 5. PMID 39182979
- [Result] Albiach-Delgado A, Moreno-Casillas JL, Ten-Domenech I, Cascant-Vilaplana MM, Moreno-Gimenez A, Gomez-Ferrer M, Sepulveda P, Kuligowski J, Quintas G. Oxylipin profile of human milk and human milk-derived extracellular vesicles. Anal Chim Acta. 2024 Jul 18;1313:342759. doi: 10.1016/j.aca.2024.342759. Epub 2024 May 21. PMID 38862207